CLINICAL TRIAL: NCT06562335
Title: Blended Therapy for Youth With a Chronic Health Condition to Increase Fatigue-related Self-efficacy (Booster): Protocol for a Multiple Baseline Single Case Experimental Study
Brief Title: The Blended Care Intervention "Booster" for Youth With Chronic Health Conditions to Increase Fatigue-related Self-efficacy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Sanne Nijhof, Principal Investigator, Pediatrician, Associate Professor, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24U-0152
Record Dates: First submitted 2024-07-24; First posted 2024-08-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Fatigue; Chronic Illnesses
Keywords: Chronic childhood disease; Fatigue; Self-efficacy; mHealth; Pediatrics; Single case
MeSH Terms: conditions — Fatigue; Chronic Disease | interventions — Immunization, Secondary

STUDY DESIGN:
Intervention Model Description: multiple baseline single case experimental AB-phase design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Booster intervention (Experimental): * Start conversation: participant personalises the Booster app, supported by the Booster practitioner
  * Measurement period: the participant fills out short repeated questionnaires 5 times daily for 4 weeks in the Booster app. This method is called experience sampling methodology (ESM). Questions are partially personalised to reflect factors that the participants believes are related to fatigue. Questions cover thoughts, feelings, and activities.
  * Insight conversation: the Booster practitioner discusses the analysed questionnaires with the participant. Together they set lifestyle goals based on the insight obtained.
  * Experiment period: the participant works on the lifestyle goals supported by the goal attainment module in the Booster app.
  Interventions: Other: Booster

INTERVENTIONS:
Other: Booster — See description of arm. The Booster intervention has evolved from the PROfeel intervention. PROfeel is described in: https://doi.org/10.1186/s13063-022-06620-2
  Other Names: PROfeel

SUMMARY:
The goal of this experimental study is to learn if the Booster intervention can be used as an early intervention for persistent fatigue. The aim of the intervention is to prevent more fatigue-related disabilities in young people with chronic illnesses like inflammatory bowel disease, childhood cancer, and juvenile idiopathic arthritis by improving self-confidence in managing fatigue (fatigue-related self-efficacy or FSE).

The main questions this study aims to answer are:

* What is the effect of the Booster intervention on fatigue-related self-efficacy (FSE)?
* What is the effect of the Booster intervention on fatigue levels, school participation, life satisfaction, and perceived health?
* When does improvement in study outcomes happen relative to the Booster intervention?
* What participant characteristics predict change in study outcomes?

Participants will follow the Booster intervention. Booster is a personalised, blended care intervention designed to help young people understand how their thoughts, feelings, and activities impact their fatigue using a smartphone app. The Booster app uses experience sampling methodology (ESM) to track these fluctuations. Based on insights obtained from these data, the participant and their healthcare provider can set personal lifestyle goals, such as increasing physical activity and reducing daytime naps. An earlier version of this intervention, called PROfeel, was effective in reducing severe fatigue. The investigators have now improved the app to also help with setting and achieving personal goals and monitoring daily progress.

The investigators will measure the effect of Booster through daily questionnaires during two phases: Phase A (baseline, before the goal setting between patient and healthcare provider) and Phase B (intervention, starting in the lifestyle change period). The duration of Phase A will be randomised for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing fatigue for at least 3 months and feeling hindered by it (Pediatric Short Fatigue Questionnaire (pSFQ) score of 15 or higher)
* Diagnosed with a chronic health condition or treated for childhood cancer

Exclusion Criteria:

Regarding other treatments:

* Fatigue fully explained by a somatic or psychiatric diagnosis
* Chronic health condition unstable in the last 3 months (e.g., recent medication changes or cancer relapse)
* Significant functional limitations due to fatigue (e.g., more than 50% school absenteeism)

Regarding feasibility:

* Cognitive impairment with an estimated IQ of below 70
* No smartphone with internet access
* Unable to speak, read, understand, or write Dutch

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue-related self-efficacy | Daily before and during the intervention, for approximately 130 days
  Single-item question, self-report via Booster app. The single item was designed and validated for this study. Answered on a VAS scale 0 to 100. Higher score represents higher fatigue-related self-efficacy.

SECONDARY OUTCOMES:
Fatigue severity | Daily before and during the intervention, for approximately 130 days
  pediatric short fatigue questionnaire, 4-item questionnaire, answered on a seven point Likert scale (1 = yes that is true, 7=no, that is not true). Total score ranges from 4 to 28, with higher scores reflecting more fatigue.
Participation | Daily before and during the intervention, for approximately 130 days
  School or work presence. Calculated: (hours present/the hours scheduled)*100
Life satisfaction | Daily before and during the intervention, for approximately 130 days
  Cantril Ladder, single-item question, rate life with ladder numbered from 0 to 10. Top of the ladder (10) represents the best possible life. The bottom (0) represents the worst possible life.
Perceived health | Daily before and during the intervention, for approximately 130 days
  EuroQol (EQ) visual analogue scale (VAS), ranging from 0 (worst health you can imagine) to 100 (best health you can imagine).

OTHER OUTCOMES:
Fatigue-related self-efficacy | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Self-Efficacy Scale-28 (SES-28) , 7-item questionnaire answered on a four-point likert scale, total scores range from 7 to 28 with higher scores indicating higher sense of control over fatigue.
Fatigue | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  PEDsQL-MFS, 23-item questionnaire
Fatigue | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Pediatric Quality of Life Inventory-Multidimensional Fatigue Scale (PEDsQL-MFS), 24-item questionnaire answered on a five-point likert (0=never, 4 = almost always), total score ranging from 0 to 96, with higher scores representing more fatigue.
Health-related quality of life | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Pediatric Quality of Life Inventory-Generic Core Scales (PEDsQL-GCS), a 23-item questionnaire answered on a five-point likert (0=never, 4 = almost always), total score ranging from 0 to 92, with higher scores representing higher quality of life. The questionnaire has the following subscales: physical, emotional, social and school or work functioning.
Health-related quality of life | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Child Health Utility Index 9D (Chu9d), nine-item questionnaire answered on a five-point likert (0 to 4), total score ranging from 0 to 36, higher scores representing lower quality of life. The Chu9D has utility values that enable calculating quality adjusted life years.
Health-related quality of life | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  EuroQol Five Dimensions Health Questionnaire Youth (EQ-5D-Y-3L), five-item questionnaire answered on a three point likert (no problems (1), some problems(2), a lot of problems(3)), total score ranging from 5 to 15, higher scores representing lower quality of life. The EQ-5D-Y-3L has utility values that enable calculating quality adjusted life years.
School or work absence | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Single item question on average absence over past half a year in %
Illness identity - fatigue | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Illness identity questionnaire (ILQ), a 25-item questionnaire, answered on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). It has the following subscales: engulfment (8 items, range 8 to 40), rejection (5 items, range 5 to 25), acceptance (5 items, range 5 to 25) and enrichment (7 items, range 7 to 35). Higher scores on subscales represent respectively higher engulfment, rejection, acceptance and enrichment. The questionnaire is adapted to specifically ask for illness identity regarding fatigue (e.g., I refuse to see my fatigue as part of myself)
Mastery | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Pearlin Schooler Mastery Scale, a seven-item questionnaire, answered on a four-point Likert scale, ranging from strongly disagree (1) to strongly agree (4). Total score ranges from 7 to 28, with higher scores reflecting higher levels of mastery.
Physical activity | Baseline, 3 months, 6 months, and if interim analysis show medium to large change also at 12 months
  Physical Activity Questionnaire for Adolescents (PAQ-A), a nine-item questionnaire. The first eight items are answered on a five-point Likert scale, ranging from low (1) to high (5) levels of physical activity. The ninth item asks whether the past week's activity was typical, less than typical, or more than typical, to provide context for the responses.The total score is calculated by averaging the scores of the first 8 items, yielding a final score ranging from 1 to 5. Higher scores indicate higher levels of physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: SL Nijhof, MSC, M.D., PhD, Principal Investigator — UMCU
Locations (1):
- Wilhelmina Children's Hospital, University Medical Centre Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Anomised individual participant data will be shared on request (see access criteria).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be avalaible after publication, and at least one year after the end of the eHealth Junior Consortium. Data remains available until the end of 2040.
Access Criteria: Participants provide consent through a consent form, specifying whether their data can be used for other research. If consent is not given, participants can still participate in the study without their data being used in these additional research contexts.
  External researchers can apply for access to data via handing in their research proposal to the principal investigator of this study. Studies concerning youth with chronic illnesses, fatigue, and studies involving extensive repeated measurements may be eligible to use the data.
  Data will be anomised before sharing to ensure privacy of participants.

REFERENCES:
- [Derived] Stutvoet MD, Vroegindeweij A, Houtveen J, van Litsenburg RRL, van de Putte E, Veltkamp RC, Nijhof SL. Blended therapy for adolescents with chronic health conditions to increase fatigue-related self-efficacy (Booster): protocol for a single-case multiple baseline study. Trials. 2025 Jul 24;26(1):255. doi: 10.1186/s13063-025-08960-1. PMID 40708017
- See also: eHealth Junior Consortium — https://ehealthjunior.nl/wordpress/